CLINICAL TRIAL: NCT07096583
Title: An Exploratory Study on NK Cell-assisted Prevention of Bone Marrow Suppression During Chemotherapy for Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Collaborators: Anhui Kecheng intelligent health technology Co., LTD (Unknown)
Responsible Party: Principal Investigator, Bai-Rong Xia, Director of Gynecological Surgery, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LLYJ-0036
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- METR-NK cell（metabolic remodeling nature killer cells） (Experimental): 100 mL METR-NK cells were diluted in 500 mL 0.9% sodium chloride normal saline at 37℃, and the infusion volume of METR-NK cells was not less than 2×107 cells/kg for 1 day as a course of treatment, and the infusion time was maintained for 30 minutes on the 10th day before chemotherapy.
  Interventions: Biological: METR-NK cell（metabolic remodeling nature killer cells）

INTERVENTIONS:
Biological: METR-NK cell（metabolic remodeling nature killer cells） — 100 mL METR-NK cells were diluted in 500 mL 0.9% sodium chloride normal saline at 37℃, and the infusion volume of METR-NK cells was not less than 2×107 cells/kg for 1 day as a course of treatment, and the infusion time was maintained for 30 minutes on the 10th day before chemotherapy.

SUMMARY:
To evaluate the remission effect and safety of intravenous injection of METR-NK cells as adjuvant therapy on bone marrow suppression in patients with ovarian cancer after chemotherapy

DETAILED DESCRIPTION:
100 mL METR-NK cells were diluted in 500 mL 0.9% sodium chloride normal saline at 37℃, and the infusion volume of METR-NK cells was not less than 2×107 cells/kg for 1 day as a course of treatment, and the infusion time was maintained for 30 minutes on the 10th day before chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old (≥18, ≤70);
* Confirmed by pathology of high grade serous ovarian cancer, high level of endometrial carcinoma, and/or primary peritoneal carcinoma fallopian tube carcinoma epithelial ovarian cancer;
* ECOG score: 0-1;
* before, during, and after treatment of blood specimen can obtain, and the participants agreed to expand blood samples to central laboratory for the trial research purposes.;
* Expectations alive at least 3 months;
* Laboratory examination indexes meet the following requirements
* (1) renal function: Cr ULN or less (upper limit of normal) x 1.5, endogenous creatinine clearance rate (Ccr) or 60 ml/min;
* (2) the liver function: the total bilirubin ULN x 1.5 or less; ALT and AST≤ULN×2.5; (If there is intrahepatic cholangiocarcinoma or liver metastasis, the total bilirubin level should be less than 3 times the upper limit of normal, and the aminotransferase level should be less than 5 times the upper limit of normal); The neutrophilic granulocyte count
* Women of childbearing age agreed to during the study and research within 6 months after the end of contraception, And non-lactating patients;
* Participants can understand the research situation and voluntarily signed informed consent. No serious complications such as active digestive tract hemorrhage, perforation, jaundice, gastrointestinal obstruction, non cancerous fever > 38 ℃;
* Expected, adherence to the good curative effect and adverse reaction will be effected according to the plan calls for follow-up

Exclusion Criteria:

* Patients had received drugs that were in other clinical trials or other cellular immunotherapies within 28 days before the screening period;
* Patients with other malignant tumours in the past five years.;
* Acute illness is ongoing, or in the past 2 years with severe disease, such as active infection, cardiovascular disease or fever patients heart function (grade III or IV level), mental health problems (such as alcohol, drugs).;
* Immunodeficiency disease, including HIV positive or suffering from other acquired and congenital immunodeficiency disease;
* Organ transplantation, organ transplantation or organ failure patients undergoing immunosuppressive medication or long-term use of immunosuppressive drugs patients;
* Move/vein thrombosis incidents happened in 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
* In patients with known to METR NK preparation any component of the final product, including the human serum albumin;
* Breastfeeding during screening serum or urine pregnancy test was positive in female;
* subjects suffering from mental illness, including major depression, mania, epilepsy, dementia, etc;
* Researchers say the other condition that doesn't fit into the group.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
The remission rate of bone marrow suppression | 3-month
  The objective of the study was to evaluate the efficacy and safety of NK cell adjuvant therapy in alleviating chemotherapy-induced myelosuppression in patients with ovarian cancer. The primary endpoints included the time to neutrophil recovery, the improvement rate of platelet count, and the incidence of infectious events

SECONDARY OUTCOMES:
Adverse event | 12-month
  Any adverse medical event that occurred after the subject received the trial drug

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospitail, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No